CLINICAL TRIAL: NCT06228859
Title: Evaluation of Locator Versus TITACH Attachment for Mandibular 2-Implant Overdentures. One-year Randomized Controlled Clinical Trial.
Brief Title: Evaluation of Locator Versus TITACH Attachment for Mandibular Overdentures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Wageh Abozaed Elsaed Mansour, Associate professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M10071020
Record Dates: First submitted 2023-12-16; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure | interventions — Denture, Overlay; Prosthodontics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (LOA): Patients were given overdentures with locator attachments. (Experimental): locater groups or overdenture attachment
  Interventions: Procedure: overdentures with different attachments
- Group II (TIA): Patients were given overdentures with TITACH attachment. (Experimental): TITACH groups for overdenture attachment
  Interventions: Procedure: overdentures with different attachments

INTERVENTIONS:
Procedure: overdentures with different attachments — different types of overdenture attachments in relation to retention, bite force, and periimplant tissue health.
  Other Names: prosthodontics

SUMMARY:
The purpose of this randomized controlled clinical study was to evaluate the locator and TITACH attachments used for retaining mandibular 2-implant overdentures regarding retention , bite force and implant marginal bone loss after overdenture insertion

DETAILED DESCRIPTION:
Locator (resilient stud) attachments have grown in favor in recent decades because they are self-aligned, give dual retention, and need less inter-arch space. The attachment's low profile may be beneficial in individuals with limited restorative space for reducing denture breakage . Furthermore, the interchangeable color-coded nylon inserts come in a variety of retention levels. Furthermore, the attachments allow for limited hinge movement and may adjust implant inclination of up to 40 degrees. However, nylon inserts exhibit significant wear and distortion and need intensive care. Elsyad et al, discovered that Locator attachments had the greatest incidence of prosthetic problems (particularly wear/distortion and replacement of retentive components) in a recent 5-year randomized controlled experiment .

A current study (TITACH) attachment (Implanova Dental Implants, Dental Evolutions Inc., USA) was designed to alleviate the issues associated with Locator attachments. Unlike the Locator system's nylon attachments, this connection enables metal-to-metal contact between the abutment and its cap. TITACH abutment, TITACH metal cap, and a silicone sleeve are the three components. When the metal cap engages the abutment, vertical holes allow it to open. The silicone sleeve functions as a block-out during cap pick-up. This type of connection may accommodate up to 33o divergence for a single implant or 66o divergence for contralateral implants. A vertical clearance of 4.5 mm and a diameter of 6 mm are required to fit the cap. It enables up to 0.2 mm of vertical cushioning, allowing for mucosal compression during function and progressive prosthesis seating. Furthermore, each attachment can withstand 7-10 lbs. of force.

Retention is the power of a dental prosthesis to withstand pressures of dislodgment along the line of installation. Prosthesis retention has been established as one of the most essential aspects in achieving successful implant overdenture therapy and increased patient satisfaction.In a previous in-vitro study, TITACH attachments were related to better retentive force results than Locator attachments, according to the authors. Although in-vitro retention testing provides for the standardization of testing conditions, Oral conditions such as mucosa, saliva, temperature, and masticatory stress may affect retention values24. Because intraoral parameters such as the presence of saliva and the structure of the residual ridge have been taken to be considered, objective assessment of clinical retention forces is preferable to subjective evaluation. Maximum biting force is determined by the activity of the jaw's elevator muscles, which is regulated by Cranio-mandibular biomechanics. In individuals with ridge resorption, dental implants will enhance biting force as part of masticatory efficiency. Mandibular implant-supported overdentures have at least double the masticatory biting force of conventional dentures.

Marginal bone loss (MBL) is a multifactorial occurrence that occurs around the cervical region of dental implants. Monitoring MBL surrounding implants is critical for determining dental implant success because it is thought to be a reliable predictor of bone response to surgery and occlusal loading. Whatever causes it, marginal bone loss is a major contributor to the development of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Complete edentulism with adequate residual alveolar bone quantity (height and width) and quality (density) at the area between the mental foramina (confirmed by cone beam CT, I -CAT, Pennsylvania, USA), 2) All patients had Angle's class I maxilla-mandibular relation with suitable inter-arch space (verified by a tentative jaw relation), and 3) All patients complained of inadequate retention and stability of their conventional mandibular dentures.

Exclusion Criteria:

* 1) systemic conditions that impede Osseo-integration, such as uncontrolled diabetes, osteoporosis, and head and neck radiation, 2) hazardous behaviors such as smoking, bruxism, and drunkenness, 3) individuals with a history of persistent TMJ disorders or reduced neuromuscular control.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Retention forces were measured using a digital force-meter. | Baseline (at time of insertion), six months, one year after insertion
  Wearing mandibular dentures and resting his chin on the apparatus chin rest, each patient was instructed to move his head until the L-shaped hooks touched the U-shaped fork at the same time. The force-meter was then moved vertically until the overdenture was removed from its position , at which point the force-meter reading in (N) was recorded. The measurements were completed three times, and the mean was calculated

SECONDARY OUTCOMES:
Maximum bite forces were measured bilaterally using a bite force transducer. | Baseline (at time of insertion), six months, one year after insertion
  The device consists of a bite fork equipped with strain gauges, which were placed between the occlusal surfaces of the denture teeth in the first molar region. Patients were instructed to bite as hard as possible on the apparatus fork for a few seconds, and measurements were taken three times for each side. Left and right force measurements were added, and the mean was statistically analyzed.

OTHER OUTCOMES:
evaluate the marginal bone loss of the dental implant for each patient. | six months and one year after insertion.
  a long cone paralleling radiographs captured by a digital device

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Wageh Abozaed, Al Mansurah, Dakahleia, Egypt